CLINICAL TRIAL: NCT06730373
Title: A Phase II, Open-Label, Multicenter Trial Comparing Disitamab Vedotin Plus Sintilimab and S-1 With Trastuzumab Plus Chemotherapy ± Sintilimab for First-Line Treatment of HER2-Positive Advanced Gastric or Gastroesophageal Junction Adenocarcinoma (RCTS2)
Brief Title: First-line Treatment With RC48 Plus Sintilimab and S-1 in Advanced Gastric Cancer (RCTS2)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Lian Liu, MD, PHD, Director, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCTS2
Record Dates: First submitted 2024-12-04; First posted 2024-12-12 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: HER2-positive Gastric Cancer; Metastatic Gastric Cancer; Unresectable Gastric Carcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — disitamab vedotin; sintilimab; S 1 (combination); Trastuzumab; Oxaliplatin; Capecitabine; Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disitamab Vedotin+Sintilimab+S-1 (Experimental)
  Interventions: Drug: Disitamab Vedotin; Drug: Sintilimab; Drug: S-1
- Trastuzumab+Chemotherapy（XELOX/FP/XP) ± Sintilimab (Active Comparator)
  Interventions: Drug: Sintilimab; Drug: Trastuzumab; Drug: Oxaliplatin; Drug: Capecitabine; Drug: 5-FU; Drug: Cisplatin

INTERVENTIONS:
Drug: Disitamab Vedotin — 2.5 mg/kg IV every 3 weeks
  Arms: Disitamab Vedotin+Sintilimab+S-1
Drug: Sintilimab — 200 mg IV every 3 weeks
Drug: S-1 — 40-60 mg BID for 14 days, every 3 weeks
  Arms: Disitamab Vedotin+Sintilimab+S-1
Drug: Trastuzumab — First load dose is 8.0mg/kg , then 6.0 mg/kg IV every 3 weeks
  Arms: Trastuzumab+Chemotherapy（XELOX/FP/XP) ± Sintilimab
Drug: Oxaliplatin — 130 mg/m2 Q3W
  Arms: Trastuzumab+Chemotherapy（XELOX/FP/XP) ± Sintilimab
Drug: Capecitabine — 1000 mg/m² Q3W
  Arms: Trastuzumab+Chemotherapy（XELOX/FP/XP) ± Sintilimab
Drug: 5-FU — 800 mg/m²
  Arms: Trastuzumab+Chemotherapy（XELOX/FP/XP) ± Sintilimab
Drug: Cisplatin — 80 mg/m²
  Arms: Trastuzumab+Chemotherapy（XELOX/FP/XP) ± Sintilimab

SUMMARY:
This is a Phase II, randomized, multicenter, open-label clinical trial designed to compare Disitamab Vedotin plus Sintilimab and S-1 with Trastuzumab plus chemotherapy ± Sintilimab for first-line treatment of HER2-Positive advanced gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged18-75 years, gender is not limited;
2. Pathologically confirmed locally advanced gastric or gastroesophageal junction adenocarcinoma that is inoperable or has distant metastasis;
3. HER2-Positive (IHC3+or IHC2+/FISH+) ;
4. Has at least 1 measurable lesion as determined by RECIST 1.1;
5. There is no systematic treatment in the past, or the patient has received neoadjuvant/adjuvant chemotherapy, but the disease progresses or relapses more than 6 months after the end of treatment;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
7. Adequate organ function;
8. The life expectancy is at least 3 months;

Exclusion Criteria:

1. Allergy to any trial drug and its excipients, or serious allergy history, or contraindication of the trial drug;
2. Cardiovascular and cerebrovascular events that are not well controlled;
3. Has received systematic treatment with Chinese patent medicine or immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use for ascites control) before the first administration within 2 weeks.
4. Have a history of interstitial lung disease, non-infectious pneumonia, pulmonary fibrosis, acute lung disease, or systemic disease with poor control (including but not limited to diabetes, hypertension, etc.);
5. Have a history of active immune deficiency or autoimmune diseases, including HIV positive test, or have other acquired or congenital immune deficiency diseases, or have a history of organ transplantation or autoimmune diseases;
6. Severe chronic or active infection requires systemic antibacterial, antifungal or antiviral treatment, including tuberculosis infection.Have a history of active tuberculosis infection ≥ 1 year before recruitment should also be excluded, unless proved has been completed appropriate treatment;
7. Brain metastasis or leptomeningeal metastasis;
8. Clinically significant pleural effusion, pericardial effusion or ascites should be drained for many times within 2 weeks before the first administration of the trial drug;
9. Has a second clinically detectable primary malignant tumor at the time of recruitment, or there were other malignant tumors in the past 5 years (except for fully treated skin basal cell carcinoma or cervical carcinoma in situ);
10. Any major surgery was performed ≤ 28 days before the first trial drug administration;
11. History of allogeneic stem cell transplantation or organ transplantation;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | 6 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) in total subjects

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 12 months after the last subject participating in
  Progression-free survival (PFS) refers to the time from the date of randomization to the first researcher's evaluation of disease progression or death (calculated by the event that occurred first). The disease progression will be evaluated by the researchers according to the RECIST 1.1 standard.
Overall survival (OS) | 12 months after the last subject participating in
  Overall survival (OS) refers to the time from the date of randomization to the date of death of the subject.
Duration of relief (DOR) | 12 months after the last subject participating in
  DOR is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death
Disease control rate (DCR) | 6 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) and stable disease(SD)in total subjects
Safety(adverse event) | Up to approximately 2 years
  to evaluate safety including adverse event rate and adverse event grade.

CONTACTS AND LOCATIONS:
Overall Officials: Lian Liu, MD, Study Chair — Qilu Hospital of Shandong University
Locations (20):
- China (20):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Shengli Oilfield Central Hospital, Dongying, Shandong
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Shandong Provincial Third Hospital, Jinan, Shandong
  - Shandong Univerisity Qilu Hospital, Jinan, Shandong
  - Jinan Third People's Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical College, Jining, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Qilu Hospital of Shandong University(Qingdao), Qingdao, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Taian City Central Hospital, Taian, Shandong
  - The Second Affiliated Hospital of Shandong First Medical University, Taian, Shandong
  - Tengzhou Central People's Hospital, Tengzhou, Shandong
  - Weifang Hospital of Traditional Chinese Medicine, Weifang, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Yantaishan Hospital, Yantai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Zibo First People's Hospital, Zibo, Shandong

IPD SHARING:
Plan to Share IPD: No